CLINICAL TRIAL: NCT03890939
Title: Effect of Servo-Ventilation on CO2 Regulation and Heart Rate Variability
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Collaborators: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASV0000001
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-01

CONDITIONS: Sleep Apnea, Mixed; Heart Failure
Keywords: Sleep Apnea, Mixed; Sleep Apnea Device; BiPap device; Sleep Study
MeSH Terms: conditions — Sleep Apnea Syndromes; Heart Failure

STUDY DESIGN:
Intervention Model Description: Participants will receive three (3) randomized PSG's during which they will receive treatment from the following devices in a randomized manner:
  * FDA released Philips BiPAP AutoSV Advanced System One
  * FDA released Philips Dreamstation BiPAP AutoSV
  * FDA released ResMed S7 VPAP Adapt
Masking Description: There will be no masking involved in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- BiPAP AutoSV Advanced System One (Experimental)
  Interventions: Device: BiPAP AutoSV Advanced System One
- Dreamstation BiPAP AutoSV (Experimental)
  Interventions: Device: Dreamstation BiPaP AutoSV
- ResMed S7 VPAP Adapt device (Active Comparator)
  Interventions: Device: ResMed S7 VPAP Adapt Device

INTERVENTIONS:
Device: BiPAP AutoSV Advanced System One — A mode of positive airway pressure used to treat sleep apnea. The difference between this device and the other experimental device is in the algorithm of the pressure settings.
  Arms: BiPAP AutoSV Advanced System One
Device: Dreamstation BiPaP AutoSV — A mode of positive airway pressure used to treat sleep apnea. The difference between this device and the other experimental device is in the algorithm of the pressure settings.
  Arms: Dreamstation BiPAP AutoSV
Device: ResMed S7 VPAP Adapt Device — A mode of positive airway pressure used to treat sleep apnea. This device is widely used by physicians to treat sleep apnea and will be the active comparator to the two experimental devices.
  Arms: ResMed S7 VPAP Adapt device

SUMMARY:
Obstructive Sleep Apnea-Hypopnea Syndrome (OSAHS) is a condition where the upper airway partially collapses and closes. This can lead to sleep problems including low oxygen levels, poor sleep, elevated carbon dioxide levels in the blood, and activation of the sympathetic nervous system. Results from having disrupted sleep may be excessive daytime sleepiness along with behavioral, functional, cardiovascular and cognitive dysfunction. Continuous Positive Airway Pressure (CPAP) is the most effective treatment for OSAHS. CPAP stabilizes the airway and prevents instability and collapse. Other forms of positive airway pressure that are approved for the treatment of OSAHS include automatically adjusting CPAP, Bi-level Positive Airway Pressure (BiPAP), and automatically adjusting BiPAP. Automatically adjusting CPAP (Auto CPAP) evaluates the airflow pattern and adjusts pressure to optimize airflow. AutoSV (Auto Servo Ventilation) is a mode of positive airway pressure used to treat obstructive and complex central sleep apnea.

In the prior study, the investigators found that the Auto S7 device led to more positive ventilation outcomes. Specifically, there was prolongation of QTc interval (the calculated time from the Q wave to the end of the T wave) and a tendency for greater premature ventricular contractions. The mechanistic basis for this could be attributable to excessive ventilation and related pro-arrhythmic effects of hypocapnia, though the investigators had not performed measures (partial pressure of CO2 (PaCO2) to detect this.

In the current study, the investigators would like to investigate the hypothesis that the S7 device leads to lower PaCO2 levels than other devices, and whether these effects are augmented in individuals with complex sleep apnea in the setting of systolic heart failure.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea-Hypopnea Syndrome (OSAHS) is a condition characterized by intermittent partial collapse and closure of the upper airway (UA). This leads to sleep fragmentation, oxygen desaturation, hypercarbia, and activation of the sympathetic nervous system. OSAHS is also associated with excessive daytime sleepiness, as well as other behavioral, functional, cardiovascular and cognitive dysfunction.

Continuous Positive Airway Pressure (CPAP) is the most effective treatment for the OSAHS. CPAP stabilizes the airway and prevents instability and collapse. With a stable airway, breathing continues in a normal manner, gas exchange is improved, and there is no disruption of sleep related to disturbed breathing.

CPAP is applied to the upper airway via a mask that covers the nose or the nose and mouth and reduces/eliminates sleep disordered breathing. The period of maximum susceptibility to airway collapse is at the end of exhalation and during early inhalation. During inhalation, negative pressures are generated in the airway by the normal process of ventilation (increase of thoracic volume and reduction of intra-thoracic pressure). The constant pressure of CPAP supports the airway throughout the ventilatory cycle.

In the sleep laboratory, titration of positive airway pressure is performed to determine effective CPAP pressures. During the procedure, the patient is instrumented for full polysomnography (PSG). Therapy is applied and pressure is adjusted during the course of the night to stabilize the upper airway and the breathing pattern. With conventional CPAP, a single pressure level is applied to the airway. While adequate for a majority of patients with obstructive sleep apnea, this static prescription will present challenges in certain patients and conditions.

Other forms of positive airway pressure that are approved for the treatment of OSAHS include automatically adjusting CPAP (Auto CPAP), Bi-level Positive Airway Pressure (BiPAP), and automatically adjusting BiPAP. Auto CPAP evaluates the airflow pattern and adjusts pressure to optimize airflow. Auto CPAP accommodates patients presenting with highly variable pressure requirements (e.g., sleep stage or body position dependent sleep apnea). The automatic adjustment can be used in patients for whom in-laboratory therapy titration is either delayed or impossible.

The REMStar Auto algorithm is proactive and flow-based. It evaluates the inspiratory flow and determines impending or actual flow limitation. This occurs in concert with a program of pressure adjustments designed to evaluate the pressure at which the airway is susceptible to collapse and maintains pressures slightly above the critical pressure. The patient is protected from "break-through" events with a full complement of intelligent responses to airflow events and snoring.

BiPAP therapy is another alternative. With BiPAP therapy, the patient's breathing pattern is monitored to identify the inspiratory and expiratory phases. Pressure is increased during inhalation and decreased during exhalation. The expiratory pressure (EPAP) is adjusted to prevent airway collapse and the inspiratory pressure (IPAP) is adjusted to prevent airflow limitation, hypopnea, snoring or arterial desaturation not associated with complete airway obstruction. BiPAP therapy differs from CPAP therapy, in that in addition to stabilizing the airway, inspiratory effort is assisted by the difference between the inspiratory and expiratory pressure.

Patients with OSAHS may be prescribed BiPAP therapy if CPAP therapy is not tolerated. BiPAP therapy may also be prescribed for patients with other respiratory disorders or for patients with both sleep and respiratory-related dysfunction.

Patients experiencing reduced ventilation from lung disease, neuromuscular disorders, or problems with the control of the breathing can experience nocturnal hypoventilation that is worse during sleep than it is during wakefulness. These patients are typically more complex and require more extensive evaluation and follow-up than patients suffering only from OSAHS. Patients may also be more vulnerable to loss or interruptions in treatment and often require more advanced modes and features such as alarms and timed back-up breaths.

OSAHS patients may respond to increases in CPAP or BiPAP therapy by demonstrating a shift in the nature of the apnea from obstructive to central. In these cases, patients may not receive adequate treatment with CPAP since lower pressure levels do not manage the instability of the airway leaving residual airway obstruction, while higher pressure levels are associated with CPAP emergent events. This condition is referred to as CPAP Emergent Complex Apnea.

Auto SV (Auto Servo Ventilation) is a mode of positive airway pressure used to treat obstructive and complex central sleep apnea. Its main features include:

* Normalization of ventilation by automatically adjusting IPAP pressure to achieve a target ventilation.
* Provision of timed, back-up breaths during central apneas. The optimal back-up rate is automatically determined by the device based on the patient's breathing.
* Automatic control of EPAP pressure to treat obstructive events.

Several manufacturers produce these types of devices. The algorithms used to determine the IPAP, EPAP and minimum respiratory rate are different. The largest number of these devices currently in use are the BiPAP AutoSV Advanced System One (Philips Respironics, Murrysville PA), Dreamstation BiPAP AutoSV and the VPAP (variable positive airway pressure) Adapt S7 (ResMed Corp., San Diego CA).

Adaptive Servo Ventilation (ASV) is a mode of positive airway pressure used to treat central sleep apnea and complex sleep apnea. The main features of the Auto SV mode include; normalization of ventilation by automatically adjusting IPAP to achieve and stabilize a target ventilation; provision of timed, back-up breaths during central apneas wherein the optimal back-up rate is automatically determined by the device based on the patient's breathing; and automatic control of EPAP to treat obstructive events.

The older version of the VPAP Adapt (S7) was found to lead to increased risk for all-cause mortality when compared to control group that involved medical management in patients with heart failure with reduced ejection fraction and predominantly central sleep apnea in a recent study (SERVE-HF). An accompanying editorial by Magalang and Pack suggested that the device algorithms may have played a role -- specifically, greater levels of pressure assist and associated increase in minute ventilation. This was supported by the measurements of minute ventilation delivered by the S7 device in the trial which was found to be greater than other servo-ventilation devices. Such increased levels of ventilation could potentially cause respiratory alkalosis which, in turn, could lead to QT interval prolongation and cardiac arrhythmias. The investigators recently performed a study of patient-ventilator interaction in patients with complex sleep apnea and preserved cardiac contractility (left ventricular ejection fraction > 45%) in order to determine the performance of various ASV devices on respiratory parameters - such as minute ventilation and apnea-hypopnea index. In order to facilitate feasibility and promote safety, the investigators avoided performing the study in the target population of the SERVE-HF trial, viz., patients with predominant central sleep apnea and heart failure with reduced ejection fraction (HFreF). The investigators performed the study only on patients with preserved ejection fraction (LVEF > 45%). In the current proposal, the investigators propose to perform the study on patients with predominantly obstructive sleep apnea and HFreF who need ASV therapy due to PAP-emergent central apneas.

In the prior study, in order to avoid intolerance to device therapy, the investigators preferred study patients who were already adherent in using servo ventilation therapy at home. The investigators will do the same in the currently proposed study. In the prior study, the investigators found that S7 device led to greater minute ventilation than other devices and that such greater levels of minute ventilation was attributable to a greater tidal volume, higher respiratory rate, and greater pressure assist. Interestingly, there was prolongation of QTc interval and a tendency for greater premature ventricular contractions in the same patients during the nights that they were exposed to the S7 device. Although the mechanistic basis for this finding is potentially attributable to excessive ventilation and related pro-arrhythmic effects of hypocapnia, the investigators had not performed measures of partial pressure of CO2 (PaCO2) in this prior study. Specifically, it is unclear whether therapy with the S7 device leads to lower PaCO2 levels than other devices and whether such effects are augmented in individuals with high loop gain (complex sleep apnea in the setting of HFreF).

Increases in minute ventilation (Ve) during wakefulness causes hypocapnia (respiratory alkalosis), which, in turn, could cause hypokalemia. Hypokalemia due to nighttime intracellular shifts in potassium ions can prolong QT interval. Conceivably, nighttime alkalosis due to excessive ventilation may lead to daytime hypokalemia and QTc prolongation through renal loss of potassium at night with consequent effects on QTc prolongation during the daytime. The observed QTc prolongation during S7 therapy was small in magnitude (~ 20 msec), but such effects may be magnified in patients with heart failure who develop metabolic alkalosis due to loop diuretics.The investigators did not, however, measure serum potassium levels which was a study limitation. In the current proposal, the investigators will ascertain the effects of nocturnal ASV therapy on serum potassium levels. Lastly, the investigators will explore the inter-individual variability in susceptibility in measured Ve or QTc interval.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide consent
* Currently prescribed servo ventilation therapy at home
* At least two weeks of recent adherence and efficacy data from PAP device demonstrating adequate use of therapy (at least 4 hours of use per night and use on at least 10 of 14 nights)
* Individuals with complex sleep apnea (obstructive sleep apnea with central apneas) and preserved left-ventricular ejection fraction (LVEF > 45%) and/or heart failure with preserved ejection fraction (HFrEF) who are currently on ASV therapy.
* Individuals with complex sleep apnea (predominantly obstructive sleep apnea with central apneas) and reduced left-ventricular ejection fraction (LVEF < 45%) and/or heart failure with reduced ejection fraction (HFrEF) who are currently on ASV therapy.

Exclusion Criteria:

* Participants who are acutely ill, medically complicated or who are medically unstable
* Participants in whom PAP therapy is otherwise medically contraindicated
* Participants who are claustrophobic
* Symptomatic ("Symptomatic" defined as hospitalized for heart failure or a change in cardiac medications, within the last two months) chronic heart failure (NYHA 2-4) AND moderate to severe predominant central sleep apnea
* Participants with previously diagnosed respiratory failure or respiratory insufficiency and who are known to have elevated arterial carbon dioxide levels while awake (PaCO2 ≥ 55mmHg).
* Participants requiring any kind of oxygen therapy
* Participants who have had surgery of the upper airway, nose, sinus, eyes, or middle ear within the previous 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Minute Ventilation | Change from Baseline through Day 4
  Minute Ventilation is the amount of air the subject moves in one minute. It is a product of the ventilatory rate and tidal volume. Scores are reported in liters per volume, and is collected from the ventilation device.
Tidal Volume | Change from Baseline through Day 4
  Tidal Volume is the lung volume representing the normal volume of air displaced between normal inhalation and exhalation when extra effort is not applied. Scores are reported in ml/kg, and is collected from the ventilation device.
Respiratory Rate | Change from Baseline through Day 4
  Respiratory Rate is measured by the number of breaths taken per minute. Scores are reported in breaths per minute, and is collected from the ventilation device.
QTc Intervals | Change from Baseline through Day 4
  QTC intervals are utilized to assess the time it takes for the heart to go from the start of the Q wave to the end of the T wave, and approximates to the time taken from when the cardiac ventricles start to contract when they finish relaxing. Scores are reported in milliseconds, and is collected from the electrocardiogram.
Acid-Base Status | Change from Baseline through Day 4
  Acid-base status is utilized to determine if subjects have increased/decreased partial carbon dioxide levels (PCO2), or decreased/increased extracellular base excess or actual Bicarbonate levels (HCO3). This is measured through transcutaneous PCO2 monitoring as well as through venipuncture blood collection. Scores are reported in millimoles per liter (mmol/l).
Electrolyte Status | Change from Baseline through Day 4
  Electrolytes Sodium (Na), Potassium (K), and Chlorine (CI) is collected through venipuncture blood collection. Scores are reported in millimoles per liter (mmol/l).

CONTACTS AND LOCATIONS:
Overall Officials: Sairam Parthasarathy, MD, Principal Investigator — University of Arizona

IPD SHARING:
Plan to Share IPD: No